CLINICAL TRIAL: NCT00128661
Title: A Double-Blind, Controlled, Randomized, Phase III Study of the Efficacy of an HPV16/18 VLP Vaccine in the Prevention of Advanced Cervical Intraepithelial Neoplasia (CIN2, CIN3, Adenocarcinoma In Situ [AIS] and Invasive Cervical Cancer) Associated With HPV 16 or HPV 18 Cervical Infection in Healthy Young Adult Women in Costa Rica.
Brief Title: Vaccine To Prevent Cervical Intraepithelial Neoplasia or Cervical Cancer in Younger Healthy Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CDR0000441189; NCI-04-C-N191; NCI-590299/009; GSK-590299/009 (Other: GSK Bio); NCT00344357 (obsolete NCT alias)
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Results first posted 2012-05-02 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-02

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical intraepithelial neoplasia grade 2; cervical cancer; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Cervarix Group (Experimental): Subjects received 3 doses of Cervarix vaccine at study Months 0, 1 and 6. All the vaccine doses were administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: human papillomavirus 16/18 L1 virus-like particle/AS04 vaccine
- Havrix Group (Active Comparator): Subjects received 3 doses of Havrix vaccine at study Months 0, 1 and 6. All the vaccine doses were administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: hepatitis A inactivated virus vaccine

INTERVENTIONS:
Biological: human papillomavirus 16/18 L1 virus-like particle/AS04 vaccine — Three doses of Cervarix vaccine administered on a 0, 1, 6-month schedule
  Arms: Cervarix Group
Biological: hepatitis A inactivated virus vaccine — Three doses of Havrix vaccine administered on a 0, 1, 6-month schedule
  Arms: Havrix Group

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer form forming, growing, or coming back. Vaccines may help the body build an effective immune response against human papillomavirus and may be effective in preventing cervical intraepithelial neoplasia or cervical cancer. It is not yet known whether human papillomavirus vaccine is more effective than hepatitis A vaccine in preventing cervical intraepithelial neoplasia or cervical cancer.

PURPOSE: This randomized phase III trial is studying human papillomavirus vaccine to see how well it works compared to hepatitis A vaccine in preventing cervical intraepithelial neoplasia or cervical cancer in younger healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

•Demonstrate the efficacy of the candidate vaccine, human papillomavirus 16/18 (HPV 16/18) L1 virus-like particle (VLP)/AS04 vaccine compared with control in preventing grade 2 or 3 cervical intraepithelial neoplasia, adenocarcinoma in situ of the cervix, or invasive cervical cancer (CIN2+) associated with HPV 16 or HPV 18 cervical infection in younger healthy participants who are negative for HPV DNA by polymerase chain reaction (PCR) for the corresponding HPV type at months 0 and 6.

Secondary

* Determine the duration of protection against HPV 16 or HPV 18 cervical infection in participants treated with the HPV 16/18 L1 VLP/AS04 vaccine.
* Determine the safety of this vaccine in these participants, regardless of their initial HPV 16/18 DNA status.
* Evaluate the efficacy of the candidate vaccine, HPV 16/18 L1 VLP/AS04 vaccine compared with control in preventing CIN2+ associated with any oncogenic HPV type cervical infection in participants who are negative for HPV DNA by PCR for the corresponding HPV type at months 0 and 6.
* Compare the efficacy of the candidate vaccine with control in preventing CIN2+ associated with HPV 16 or HPV 18 cervical infection, detected within the lesional component of the cervical tissue specimen by PCR, in participants who are negative for HPV DNA by PCR for the corresponding HPV type at months 0 and 6 and by enzyme-linked immunosorbent assay (ELISA) at month 0.
* Compare the efficacy of the candidate vaccine with control in preventing persistent HPV 16 or HPV 18 cervical infection in these participants.
* Determine the immunogenicity of HPV 16/18 L1 VLP/AS04 vaccine by ELISA and V5/J4 monoclonal antibody inhibition enzyme immunoassay in the first 600 participants randomized to receive HPV 16/18 L1 VLP/AS04 vaccine.

OUTLINE: This is a randomized, controlled, double-blind, parallel-group study. Participants are randomized to 1 of 2 treatment arms.

* Arm I: Participants receive human papillomavirus 16/18 L1 virus-like particle/AS04 vaccine intramuscularly (IM) once in months 0, 1, and 6.
* Arm II: Participants receive hepatitis A vaccine (Havrix®) IM once in months 0, 1, and 6.

After completion of study treatment, participants are followed at 6 months and then at least annually for 3 years.

PROJECTED ACCRUAL: Approximately 7,500 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

•Healthy participants

* Deemed to be in good general health by history and physical examination

  •Resident of Guanacaste Province of Costa Rica and surrounding areas
* Must remain a resident for ≥ 6 months after the first study vaccination

PATIENT CHARACTERISTICS:

Age

* 18 to 25

Performance status

•Not specified

Life expectancy

•Not specified

Hematopoietic

•Not specified

Hepatic

* No history of chronic hepatitis requiring treatment
* No acute or chronic clinically significant hepatic function abnormality by physical examination or laboratory findings
* No known history of hepatitis A infection

Renal

* No history of kidney disease requiring treatment
* No acute or chronic clinically significant kidney function abnormality by physical examination or laboratory findings

Cardiovascular

* No acute or chronic clinically significant cardiovascular function abnormality by physical examination or laboratory findings Pulmonary
* No acute or chronic clinically significant pulmonary function abnormality by physical examination or laboratory findings Immunology
* No history of allergic disease
* No history of autoimmune disorder requiring treatment
* No history of allergic reaction (e.g., difficulty breathing) to any vaccine
* No suspected allergy or reaction likely to be exacerbated by a component of the study vaccines (e.g., 2-phenoxyethanol or neomycin)
* No hypersensitivity to latex
* No diagnosis or suspicion of any immunodeficient condition by medical history or physical examination Other
* Not pregnant or nursing

  ◦No delivery within the past 3 months
* Negative pregnancy test
* Fertile patients must use effective contraception for 30 days before, during, and for 60 days after completion of study treatment
* Able to speak or understand Spanish
* Mentally competent
* Able to undergo pelvic exam (i.e., no heavy bleeding [menstruation or otherwise] or heavy vaginal discharge)
* No history of cancer requiring treatment
* No history of diabetes requiring treatment
* No history of other chronic conditions requiring treatment
* No acute or chronic clinically significant neurologic function abnormality by physical examination or laboratory findings
* No other acute disease
* No fever ≥ 37.5º C

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 6 months since prior chronic administration (i.e., > 14 days) of immune-modulating drugs
* More than 90 days since prior immunoglobulins
* More than 30 days since prior and no other concurrent investigational or non-registered vaccines
* More than 30 days since prior registered vaccines
* More than 8 days since prior routine meningococcal, hepatitis B, influenza, or diphtheria/tetanus vaccine
* No prior vaccination against hepatitis A
* No prior vaccination against human papillomavirus
* No prior monophosphoryl lipid A or AS04 adjuvant

Chemotherapy

•Not specified

Endocrine therapy

* More than 6 months since prior chronic administration (i.e., > 14 days) of corticosteroids (e.g., ≥ 0.5 mg/kg/day of prednisone or equivalent)
* Concurrent inhaled or topical steroids allowed

Radiotherapy

•Not specified

Surgery

•No prior hysterectomy

Other

* More than 6 months since prior chronic administration (i.e., > 14 days) of immunosuppressants
* More than 30 days since prior and no other concurrent investigational or non-registered drugs

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7466 (Actual)
Dates: Start 2004-06-30 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2010-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Proyecto Epidemiologico Guanacaste, Liberia, Costa Rica

REFERENCES:
- [Background] Kreimer AR, Rodriguez AC, Hildesheim A, Herrero R, Porras C, Schiffman M, Gonzalez P, Solomon D, Jimenez S, Schiller JT, Lowy DR, Quint W, Sherman ME, Schussler J, Wacholder S; CVT Vaccine Group. Proof-of-principle evaluation of the efficacy of fewer than three doses of a bivalent HPV16/18 vaccine. J Natl Cancer Inst. 2011 Oct 5;103(19):1444-51. doi: 10.1093/jnci/djr319. Epub 2011 Sep 9. PMID 21908768
- [Background] Kemp TJ, Hildesheim A, Safaeian M, Dauner JG, Pan Y, Porras C, Schiller JT, Lowy DR, Herrero R, Pinto LA. HPV16/18 L1 VLP vaccine induces cross-neutralizing antibodies that may mediate cross-protection. Vaccine. 2011 Mar 3;29(11):2011-4. doi: 10.1016/j.vaccine.2011.01.001. Epub 2011 Jan 15. PMID 21241731
- [Derived] Sierra MS, Coto C, Porras C, Herrero R, Ugalde D, Sauer AN, Mora D, Montes CP, Schussler J, Hoffman AC, Hicks B, Ruggieri D, Cortes B, Hildesheim A, Kreimer AR, Wentzensen N, Dagnall C, Liu D. Validation of TypeSeq2, a Next-Generation-Based Sequencing Assay for the Detection of 46 Human Papillomavirus Genotypes, at the US National Cancer Institute and Costa Rica Laboratories. J Infect Dis. 2025 Dec 20;232(6):e906-e915. doi: 10.1093/infdis/jiaf369. PMID 40796225
- [Derived] Sierra MS, Carvajal LJ, Dull P, Herrero R, Schussler J, Hildesheim A, Schiller JT, Ocampo R, Liu D, Kreimer AR, Rodriguez AC, Lowy DR, Porras C; Costa Rica HPV Vaccine Trial (CVT) Group. Human papillomavirus type 16 and 18 viral clearance and progression to precancer among women aged 18-25 years enrolled in the Costa Rica HPV prophylactic vaccine trial (CVT). Vaccine. 2025 Mar 19;50:126841. doi: 10.1016/j.vaccine.2025.126841. Epub 2025 Feb 16. PMID 39961279
- [Derived] Befano B, Campos NG, Egemen D, Herrero R, Schiffman M, Porras C, Lowy DR, Rodriguez AC, Schiller JT, Ocampo R, Hildesheim A, Sampson JN, Das S, Kreimer AR, Cheung LC; Costa Rica HPV Vaccine Trial (CVT) Group. Estimating human papillomavirus vaccine efficacy from a single-arm trial: proof-of-principle in the Costa Rica Vaccine Trial. J Natl Cancer Inst. 2023 Jul 6;115(7):788-795. doi: 10.1093/jnci/djad064. PMID 37040086
- [Derived] Sierra MS, Tsang SH, Porras C, Herrero R, Sampson JN, Cortes B, Schussler J, Wagner S, Carvajal L, Quint W, Kreimer AR, Hu S, Rodriguez AC, Romero B, Hildesheim A; Costa Rica HPV Vaccine Trial (CVT) Group. Analysis of cervical HPV infections among unvaccinated young adult women to inform vaccine strategies in this age group: the Costa Rica HPV Vaccine Trial. Sex Transm Infect. 2022 Jul 16;99(3):180-6. doi: 10.1136/sextrans-2022-055434. Online ahead of print. PMID 35842229
- [Derived] Shing JZ, Hu S, Herrero R, Hildesheim A, Porras C, Sampson JN, Schussler J, Schiller JT, Lowy DR, Sierra MS, Carvajal L, Kreimer AR; Costa Rica HPV Vaccine Trial Group. Precancerous cervical lesions caused by non-vaccine-preventable HPV types after vaccination with the bivalent AS04-adjuvanted HPV vaccine: an analysis of the long-term follow-up study from the randomised Costa Rica HPV Vaccine Trial. Lancet Oncol. 2022 Jul;23(7):940-949. doi: 10.1016/S1470-2045(22)00291-1. Epub 2022 Jun 13. PMID 35709811
- [Derived] Usyk M, Schlecht NF, Pickering S, Williams L, Sollecito CC, Gradissimo A, Porras C, Safaeian M, Pinto L, Herrero R, Strickler HD, Viswanathan S, Nucci-Sack A, Diaz A; Costa Rica HPV Vaccine Trial (CVT) Group; Burk RD. molBV reveals immune landscape of bacterial vaginosis and predicts human papillomavirus infection natural history. Nat Commun. 2022 Jan 11;13(1):233. doi: 10.1038/s41467-021-27628-3. PMID 35017496
- [Derived] Usyk M, Zolnik CP, Castle PE, Porras C, Herrero R, Gradissimo A, Gonzalez P, Safaeian M, Schiffman M, Burk RD; Costa Rica HPV Vaccine Trial (CVT) Group. Cervicovaginal microbiome and natural history of HPV in a longitudinal study. PLoS Pathog. 2020 Mar 26;16(3):e1008376. doi: 10.1371/journal.ppat.1008376. eCollection 2020 Mar. PMID 32214382
- [Derived] Safaeian M, Castellsague X, Hildesheim A, Wacholder S, Schiffman MH, Bozonnat MC, Baril L, Rosillon D; Costa Rica HPV Vaccine Trial and the PATRICIA study groups. Risk of HPV-16/18 Infections and Associated Cervical Abnormalities in Women Seropositive for Naturally Acquired Antibodies: Pooled Analysis Based on Control Arms of Two Large Clinical Trials. J Infect Dis. 2018 Jun 5;218(1):84-94. doi: 10.1093/infdis/jiy112. PMID 29718393
- [Derived] Hildesheim A, Gonzalez P, Kreimer AR, Wacholder S, Schussler J, Rodriguez AC, Porras C, Schiffman M, Sidawy M, Schiller JT, Lowy DR, Herrero R; Costa Rica HPV Vaccine Trial (CVT) Group. Impact of human papillomavirus (HPV) 16 and 18 vaccination on prevalent infections and rates of cervical lesions after excisional treatment. Am J Obstet Gynecol. 2016 Aug;215(2):212.e1-212.e15. doi: 10.1016/j.ajog.2016.02.021. Epub 2016 Feb 16. PMID 26892991
- [Derived] Beachler DC, Kreimer AR, Schiffman M, Herrero R, Wacholder S, Rodriguez AC, Lowy DR, Porras C, Schiller JT, Quint W, Jimenez S, Safaeian M, Struijk L, Schussler J, Hildesheim A, Gonzalez P; Costa Rica HPV Vaccine Trial (CVT) Group. Multisite HPV16/18 Vaccine Efficacy Against Cervical, Anal, and Oral HPV Infection. J Natl Cancer Inst. 2015 Oct 14;108(1):djv302. doi: 10.1093/jnci/djv302. Print 2016 Jan. PMID 26467666
- [Derived] Panagiotou OA, Befano BL, Gonzalez P, Rodriguez AC, Herrero R, Schiller JT, Kreimer AR, Schiffman M, Hildesheim A, Wilcox AJ, Wacholder S; Costa Rica HPV Vaccine Trial (CVT) Group (see end of manuscript for full list of investigators). Effect of bivalent human papillomavirus vaccination on pregnancy outcomes: long term observational follow-up in the Costa Rica HPV Vaccine Trial. BMJ. 2015 Sep 7;351:h4358. doi: 10.1136/bmj.h4358. PMID 26346155
- [Derived] Kreimer AR, Struyf F, Del Rosario-Raymundo MR, Hildesheim A, Skinner SR, Wacholder S, Garland SM, Herrero R, David MP, Wheeler CM; Costa Rica Vaccine Trial Study Group Authors; Gonzalez P, Jimenez S, Lowy DR, Pinto LA, Porras C, Rodriguez AC, Safaeian M, Schiffman M, Schiller JT, Schussler J, Sherman ME; PATRICIA Study Group Authors; Bosch FX, Castellsague X, Chatterjee A, Chow SN, Descamps D, Diaz-Mitoma F, Dubin G, Germar MJ, Harper DM, Lewis DJ, Limson G, Naud P, Peters K, Poppe WA, Ramjattan B, Romanowski B, Salmeron J, Schwarz TF, Teixeira JC, Tjalma WA; HPV PATRICIA Principal Investigators/Co-Principal Investigator Collaborators; GSK Vaccines Clinical Study Support Group. Efficacy of fewer than three doses of an HPV-16/18 AS04-adjuvanted vaccine: combined analysis of data from the Costa Rica Vaccine and PATRICIA Trials. Lancet Oncol. 2015 Jul;16(7):775-86. doi: 10.1016/S1470-2045(15)00047-9. Epub 2015 Jun 9. PMID 26071347
- [Derived] Gonzalez P, Hildesheim A, Herrero R, Katki H, Wacholder S, Porras C, Safaeian M, Jimenez S, Darragh TM, Cortes B, Befano B, Schiffman M, Carvajal L, Palefsky J, Schiller J, Ocampo R, Schussler J, Lowy D, Guillen D, Stoler MH, Quint W, Morales J, Avila C, Rodriguez AC, Kreimer AR; Costa Rica HPV Vaccine Trial (CVT) Group. Rationale and design of a long term follow-up study of women who did and did not receive HPV 16/18 vaccination in Guanacaste, Costa Rica. Vaccine. 2015 Apr 27;33(18):2141-51. doi: 10.1016/j.vaccine.2015.03.015. Epub 2015 Mar 18. PMID 25796338
- [Derived] Lang Kuhs KA, Porras C, Schiller JT, Rodriguez AC, Schiffman M, Gonzalez P, Wacholder S, Ghosh A, Li Y, Lowy DR, Kreimer AR, Poncelet S, Schussler J, Quint W, van Doorn LJ, Sherman ME, Sidawy M, Herrero R, Hildesheim A, Safaeian M; Costa Rica Vaccine Trial Group. Effect of different human papillomavirus serological and DNA criteria on vaccine efficacy estimates. Am J Epidemiol. 2014 Sep 15;180(6):599-607. doi: 10.1093/aje/kwu168. Epub 2014 Aug 19. PMID 25139208
- [Derived] Hildesheim A, Wacholder S, Catteau G, Struyf F, Dubin G, Herrero R; CVT Group. Efficacy of the HPV-16/18 vaccine: final according to protocol results from the blinded phase of the randomized Costa Rica HPV-16/18 vaccine trial. Vaccine. 2014 Sep 3;32(39):5087-97. doi: 10.1016/j.vaccine.2014.06.038. Epub 2014 Jul 10. PMID 25018097
- [Derived] Lang Kuhs KA, Gonzalez P, Rodriguez AC, van Doorn LJ, Schiffman M, Struijk L, Chen S, Quint W, Lowy DR, Porras C, DelVecchio C, Jimenez S, Safaeian M, Schiller JT, Wacholder S, Herrero R, Hildesheim A, Kreimer AR; Costa Rica Vaccine Trial Group. Reduced prevalence of vulvar HPV16/18 infection among women who received the HPV16/18 bivalent vaccine: a nested analysis within the Costa Rica Vaccine Trial. J Infect Dis. 2014 Dec 15;210(12):1890-9. doi: 10.1093/infdis/jiu357. Epub 2014 Jun 23. PMID 24958910
- [Derived] Lang Kuhs KA, Gonzalez P, Struijk L, Castro F, Hildesheim A, van Doorn LJ, Rodriguez AC, Schiffman M, Quint W, Lowy DR, Porras C, Delvecchio C, Katki HA, Jimenez S, Safaeian M, Schiller J, Solomon D, Wacholder S, Herrero R, Kreimer AR; Costa Rica Vaccine Trial Group. Prevalence of and risk factors for oral human papillomavirus among young women in Costa Rica. J Infect Dis. 2013 Nov 15;208(10):1643-52. doi: 10.1093/infdis/jit369. Epub 2013 Sep 6. PMID 24014882
- [Derived] Herrero R, Quint W, Hildesheim A, Gonzalez P, Struijk L, Katki HA, Porras C, Schiffman M, Rodriguez AC, Solomon D, Jimenez S, Schiller JT, Lowy DR, van Doorn LJ, Wacholder S, Kreimer AR; CVT Vaccine Group. Reduced prevalence of oral human papillomavirus (HPV) 4 years after bivalent HPV vaccination in a randomized clinical trial in Costa Rica. PLoS One. 2013 Jul 17;8(7):e68329. doi: 10.1371/journal.pone.0068329. Print 2013. PMID 23873171
- [Derived] Clarke M, Schiffman M, Wacholder S, Rodriguez AC, Hildesheim A, Quint W; Costa Rican Vaccine Trial Group. A prospective study of absolute risk and determinants of human papillomavirus incidence among young women in Costa Rica. BMC Infect Dis. 2013 Jul 8;13:308. doi: 10.1186/1471-2334-13-308. PMID 23834901
- [Derived] Castro FA, Quint W, Gonzalez P, Katki HA, Herrero R, van Doorn LJ, Schiffman M, Struijk L, Rodriguez AC, DelVecchio C, Lowy DR, Porras C, Jimenez S, Schiller J, Solomon D, Wacholder S, Hildesheim A, Kreimer AR; Costa Rica Vaccine Trial Group. Prevalence of and risk factors for anal human papillomavirus infection among young healthy women in Costa Rica. J Infect Dis. 2012 Oct 1;206(7):1103-10. doi: 10.1093/infdis/jis458. Epub 2012 Jul 30. PMID 22850119
- [Derived] Kreimer AR, Gonzalez P, Katki HA, Porras C, Schiffman M, Rodriguez AC, Solomon D, Jimenez S, Schiller JT, Lowy DR, van Doorn LJ, Struijk L, Quint W, Chen S, Wacholder S, Hildesheim A, Herrero R; CVT Vaccine Group. Efficacy of a bivalent HPV 16/18 vaccine against anal HPV 16/18 infection among young women: a nested analysis within the Costa Rica Vaccine Trial. Lancet Oncol. 2011 Sep;12(9):862-70. doi: 10.1016/S1470-2045(11)70213-3. Epub 2011 Aug 22. PMID 21865087
- [Derived] Wacholder S, Chen BE, Wilcox A, Macones G, Gonzalez P, Befano B, Hildesheim A, Rodriguez AC, Solomon D, Herrero R, Schiffman M; CVT group. Risk of miscarriage with bivalent vaccine against human papillomavirus (HPV) types 16 and 18: pooled analysis of two randomised controlled trials. BMJ. 2010 Mar 2;340:c712. doi: 10.1136/bmj.c712. PMID 20197322
- [Derived] Dessy FJ, Giannini SL, Bougelet CA, Kemp TJ, David MP, Poncelet SM, Pinto LA, Wettendorff MA. Correlation between direct ELISA, single epitope-based inhibition ELISA and pseudovirion-based neutralization assay for measuring anti-HPV-16 and anti-HPV-18 antibody response after vaccination with the AS04-adjuvanted HPV-16/18 cervical cancer vaccine. Hum Vaccin. 2008 Nov-Dec;4(6):425-34. doi: 10.4161/hv.4.6.6912. Epub 2008 Nov 11. PMID 18948732
- [Derived] Hildesheim A, Herrero R, Wacholder S, Rodriguez AC, Solomon D, Bratti MC, Schiller JT, Gonzalez P, Dubin G, Porras C, Jimenez SE, Lowy DR; Costa Rican HPV Vaccine Trial Group. Effect of human papillomavirus 16/18 L1 viruslike particle vaccine among young women with preexisting infection: a randomized trial. JAMA. 2007 Aug 15;298(7):743-53. doi: 10.1001/jama.298.7.743. PMID 17699008

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Solicited symptoms were collected for 3730 and 3740 subjects instead of the 3727 and 3739 subjects who were randomized in the study in the Cervarix and the Havrix groups, respectively. These 4 subjects received both vaccines and were included in the denominator of both arm based on the actual vaccine type administered.
Period: Overall Study
Arm/Group | Cervarix Group | Havrix Group
Started | 3727 | 3739
Completed | 3453 | 3481
Not Completed | 274 | 258
Not completed — Adverse Event | 14 | 11
Not completed — Lost to Follow-up | 10 | 7
Not completed — Withdrawal by Subject | 243 | 232
Not completed — Other | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Havrix Group | Total
Number analyzed (Participants) | 3727 | 3739 | 7466
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Years | 21.1 (2.3) | 21.1 (2.3) | 21.1 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3727 | 3739 | 7466
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Histopathologically Confirmed Cervical Intraepithelial Neoplasia (CIN)2+ Cases Associated With HPV16 and/or HPV18 Infection Detected in the Preceding Cervical Cytology Specimen.
Description: CIN2+ was defined as CIN grade 2 (CIN2), CIN grade 3 (CIN3), adenocarcinoma in situ (AIS) or invasive cervical cancer. Preceding cervical cytology means the last cervical cytology specimen collected before the histopathology specimen was obtained. Subjects were human papillomavirus (HPV) deoxyribonucleic acid (DNA) negative (DNA-) by polymerase chain reaction (PCR) at Month 0 and Month 6 for the corresponding HPV-type.
Time Frame: From Month 6 up to Month 48
Population: The According-To-Protocol (ATP) cohort for efficacy included subjects with efficacy data available, who received 3 doses of vaccine, who were HPV DNA- for the corresponding type at enrollment and at the time of administration of the 3rd dose (Month 6) and who did not have a biopsy or treatment during the vaccination phase (prior to the Month 6).
Measure: Number; unit: Events
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 2635 | 2677
Events
  HPV16 Associated CIN2+ (N=2464;2452) | 1 | 9
  HPV18 Associated CIN2+ (N=2567; 2593) | 0 | 2
  HPV16 and/or 18 Associated CIN2+ (N=2635;2677) | 1 | 10

2. Secondary Outcome: Number of Cervical Infection With HPV16 or HPV18.
Description: Subjects were human papillomavirus (HPV) deoxyribonucleic acid (DNA) negative (DNA-) (by PCR) at Month 0 and Month 6 for the corresponding HPV-type
Time Frame: From Month 6 up to Month 48
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 2635 | 2677
Events
  HPV16 Cervical Infection (N=2464;2452) | 50 | 251
  HPV18 Cervical Infection (N=2567;2593) | 32 | 177
  HPV16 and/or 18 Cervical Infection (N=2635;2677) | 78 | 387

3. Secondary Outcome: Number of Histopathologically Confirmed CIN2+ Cases Associated With Infection by Any Oncogenic HPV Type
Description: Oncogenic HPV types included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59 and 68 detected by polymerase chain reaction (PRC) in the preceding cervical cytology specimen. Note: The assay did not distinguish between HPV types 68 and 73. CIN2+ was defined as CIN grade 2 (CIN2), CIN grade 3 (CIN3), adenocarcinoma in situ (AIS) or invasive cervical cancer Subjects were human papillomavirus (HPV) deoxyribonucleic acid (DNA) negative (DNA-) (by PCR) at Month 0 and Month 6 for the corresponding HPV-type
Time Frame: From Month 6 up to Month 48
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 2643 | 2697
Events
  HPV16 Associated CIN2+ (N=2464;2452) | 1 | 9
  HPV18 Associated CIN2+ (N=2567,2593) | 0 | 2
  HPV31 Associated CIN2+ (N=2525;2546) | 1 | 6
  HPV33 Associated CIN2+ (N=2596;2645) | 0 | 3
  HPV35 Associated CIN2+ (N=2593;2631) | 0 | 4
  HPV39 Associated CIN2+ (N=2528;2581) | 0 | 0
  HPV45 Associated CIN2+ (N=2573;2622) | 1 | 1
  HPV51 Associated CIN2+ (N=2453;2539) | 1 | 6
  HPV52 Associated CIN2+ (N=2456;2505) | 5 | 10
  HPV56 Associated CIN2+ (N=2524;2564) | 1 | 5
  HPV58 Associated CIN2+ (N=2551;2595) | 2 | 5
  HPV59 Associated CIN2+ (N=2576;2637) | 3 | 3
  HPV68 and/or 73 Associated CIN2+ (N=2519;2576) | 1 | 4
  Non 16/18 Onco HPV Associated CIN2+ (N=2643;2697) | 11 | 28
  Any Oncogenic HPV Associated CIN2+ (N=2643;2697) | 11 | 33

4. Secondary Outcome: Number of Persistent Infection (12-month Definition) With Human Papillomavirus (HPV)-16 or HPV-18 Cases
Description: Persistent incident HPV-16 and /or HPV-18 cervical infection had to fulfil the following criteria: first detection after the 6-month visit, 2 same type HPV positive (by PCR) test results 10+ months apart, and no intervening HPV negative tests for the corresponding type. Persistent HPV16 or HPV18 cervical infection = detection of the same HPV type by polymerase chain reaction (PCR) in cervical samples from all consecutive evaluations over approximately 12 months. Subjects were HPV deoxyribonucleic acid (DNA) negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type.
Time Frame: From Month 6 up to Month 48
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 2635 | 2677
Events
  Persistent HPV16 Infection (N=2464,2452) | 10 | 71
  Persistent HPV18 Infection (N=2567;2593) | 0 | 37
  Persistent HPV16 and/or 18 Infection (N=2635;2677) | 10 | 104

5. Secondary Outcome: Geometric Mean Titers (GMTs) for HPV-16 Antibody in the Immunogenicity Subcohort.
Description: Titers were assessed for the 600 subjects enrolled into the immunogenicity subcohort by Enzyme linked immunosorbent assay (ELISA) and expressed as geometric mean titers (GMTs). Seronegative subjects = antibody concentration below 8 ELISA Units per millilitre (EL.U/mL) prior to vaccination. Seropositive subjects=antibody concentration equal to or above 8 EL.U/mL prior to vaccination. Immunogenicity subcohort = subset of 600 subjects from the 2 groups of the ATP cohort: subjects attended 1 extra clinic visit approximately 1 month (30 to 60 days) after the last dose was administered (Month 7)
Time Frame: Before vaccination and at Month 1, 6, 7, 12, 18, 24, 30, 36, 42 and 48
Population: The ATP cohort for immunogenicity included subjects who received 3 doses of vaccine, who were HPV DNA- for the corresponding type at enrollment and during the 48-month follow-up period, who did not have a biopsy or treatment during the vaccination phase (prior to the Month 6) and for whom immunogenicity results were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 196 | 157
Titers
  HPV-16 [before vaccination] (N=194;156) | 6.7 [5.7 to 7.8] | 8.2 [6.7 to 10.0]
  HPV-16 [at Month 1] (N=196,157) | 646.6 [549.3 to 761.1] | 7.9 [6.5 to 9.6]
  HPV-16 [at Month 6] (N=195,156) | 771.5 [668.3 to 890.7] | 8.4 [6.9 to 10.3]
  HPV-16 [at Month 7] (N=195,157) | 3261 [2959 to 3595] | 8.5 [6.9 to 10.3]
  HPV-16 [at Month 12] (N=182,146) | 2090 [1822 to 2398] | 8.3 [6.7 to 10.4]
  HPV-16 [at Month 18] (N=25,17) | 1045 [776.0 to 1408] | 10.4 [4.8 to 22.7]
  HPV-16 [at Month 24] (N=175,137) | 1486 [1293 to 1709] | 8.6 [6.9 to 10.7]
  HPV-16 [at Month 30] (N=19,15) | 1070 [747.5 to 1532] | 11.9 [5.1 to 28.0]
  HPV-16 [at Month 36] (N=163,132) | 1256 [1080 to 1461] | 9.0 [7.4 to 11.0]
  HPV-16 [at Month 42] (N=22,18) | 1259 [879.4 to 1802] | 6.1 [4.0 to 9.4]
  HPV-16 [at Month 48] (N=172,131) | 1155 [1009 to 1322] | 9.5 [7.7 to 11.7]

6. Secondary Outcome: Geometric Mean Titers (GMTs) for HPV-18 Antibody in the Immunogenicity Subcohort
Description: Titers were assessed for the 600 subjects enrolled into the immunogenicity subcohortby Enzyme linked immunosorbent assay (ELISA) and expressed as geometric mean titers (GMTs). Seronegative (Sero-) subjects=antibody concentration below 7 EL.U/mL prior to vaccination. Seropositive (Sero+) subjects=antibody concentration equal to or above 7 EL.U/mL prior to vaccination. Immunogenicity subcohort=subset of 600 subjects from the 2 groups of the ATP cohort: subjects attended 1 extra clinic visit approximately 1 month (30 to 60 days) after the last dose was administered (Month 7).
Time Frame: Before vaccination and at Month 1, 6, 7, 12, 18, 24, 30, 36, 42 and 48
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 203 | 175
Titers
  HPV-18 [before vaccination] (N=200;173) | 5.4 [4.8 to 6.1] | 6.2 [5.2 to 7.4]
  HPV-18 [at Month 1] (N=203;170) | 372.7 [322.8 to 430.3] | 6.4 [5.4 to 7.6]
  HPV-18 [at Month 6] (N=203;175) | 532.2 [467.5 to 605.9] | 6.7 [5.6 to 7.9]
  HPV-18 [at Month 7] (N=202;175) | 3276 [3001 to 3576] | 6.8 [5.7 to 8.1]
  HPV-18 [at Month 12] (N=190;166) | 1082 [942.0 to 1242] | 7.0 [5.7 to 8.5]
  HPV-18 [at Month 18] (N=28;20) | 502.4 [339.1 to 744.5] | 6.7 [3.8 to 12.1]
  HPV-18 [at Month 24] (N=178;150) | 633.0 [551.5 to 726.6] | 6.9 [5.6 to 8.4]
  HPV-18 [at Month 30] (N=17;19) | 403.8 [257.8 to 632.5] | 6.4 [3.8 to 10.5]
  HPV-18 [at Month 36] (N=168;145) | 519.7 [449.3 to 601.1] | 6.0 [5.0 to 7.2]
  HPV-18 [at Month 42] (N=25;19) | 582.4 [422.9 to 801.9] | 5.5 [3.6 to 8.4]
  HPV-18 [at Month 48] (N=179;149) | 470.1 [411.2 to 537.4] | 6.6 [5.5 to 8.0]

7. Secondary Outcome: HPV-16 Geometric Mean Titers (GMTs) (V5 Monoclonal Antibody Inhibition Test)
Description: Titers were assessed for the 600 subjects enrolled into the immunogenicity subcohort by Inhibition Enzyme Immunoassay (EIA) and expressed as geometric mean antibody titers (GMTs). Seronegative (Sero-) subjects=antibody concentration below 41 EL.U/mL prior to vaccination. Seropositive (Sero+) subjects=antibody concentration equal to or above 41 EL.U/mL prior to vaccination. Immunogenicity subcohort=subset of 600 subjects from the 2 groups of the ATP cohort: subjects attended 1 extra clinic visit approximately 1 month (30 to 60 days) after the last dose was administered (Month 7).
Time Frame: Before vaccination and at Month 1, 6, 7, 12, 18, 24, 30, 36, 42 and 48
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 196 | 158
Titers
  HPV-16 [before vaccination] (N=196;158) | 21.1 [20.5 to 21.8] | 21.4 [20.6 to 22.3]
  HPV-16 [at Month 1] (N=182;155) | 58.5 [48.3 to 70.8] | 21.5 [20.7 to 22.3]
  HPV-16 [at Month 6] (N=189;156) | 80.9 [70.3 to 93.1] | 21.5 [20.6 to 22.4]
  HPV-16 [at Month 7] (N=193;158) | 1047 [926.3 to 1183] | 21.4 [20.6 to 22.3]
  HPV-16 [at Month 12] (N=175;146) | 291.4 [253.7 to 334.8] | 22.6 [20.8 to 24.5]
  HPV-16 [at Month 18] (N=24;17) | 116.6 [83.2 to 163.3] | 20.5 [20.5 to 20.5]
  HPV-16 [at Month 24] (N=169;138) | 184.6 [163.0 to 209.1] | 21.4 [20.6 to 22.3]
  HPV-16 [at Month 30] (N=18;15) | 112.4 [78.7 to 160.6] | 20.5 [20.5 to 20.5]
  HPV-16 [at Month 36] (N=162;132) | 139.7 [122.5 to 159.5] | 20.8 [20.2 to 21.3]
  HPV-16 [at Month 42] (N=22;18) | 126.9 [89.9 to 179.1] | 20.5 [20.5 to 20.5]
  HPV-16 [at Month 48] (N=168;133) | 131.8 [115.5 to 150.5] | 21.0 [20.4 to 21.7]

8. Secondary Outcome: HPV-18 Geometric Mean Titers (GMTs) (J4 Monoclonal Antibody Inhibition Test)
Description: Titers were assessed for the 600 subjects enrolled into the immunogenicity subcohort by Inhibition Enzyme Immunoassay (EIA) and expressed as geometric mean antibody titers (GMTs). Seronegative (Sero-) subjects=antibody concentration below 110 EL.U/mL prior to vaccination. Seropositive (Sero+) subjects=antibody concentration equal to or above 110 EL.U/mL prior to vaccination. Immunogenicity subcohort=subset of 600 subjects from the 2 groups of the ATP cohort: subjects attended 1 extra clinic visit approximately 1 month (30 to 60 days) after the last dose was administered (Month 7).
Time Frame: Before vaccination and at Month 1, 6, 7, 12, 18, 24, 30, 36, 42 and 48
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 203 | 176
Titers
  HPV-18 [before vaccination] (N=203;176) | 55.0 [55.0 to 55.0] | 55.7 [54.7 to 56.7]
  HPV-18 [at Month 1] (N=197;173) | 99.1 [88.0 to 111.5] | 55.3 [54.7 to 55.8]
  HPV-18 [at Month 6] (N=195;175) | 111.4 [100.2 to 123.9] | 55.4 [54.6 to 56.3]
  HPV-18 [at Month 7] (N=198;176) | 823.6 [737.7 to 919.5] | 55.0 [55.0 to 55.0]
  HPV-18 [at Month 12] (N=182;166) | 231.1 [203.2 to 262.7] | 56.7 [54.7 to 58.8]
  HPV-18 [at Month 18] (N=28;20) | 121.8 [89.5 to 165.8] | 55.0 [55.0 to 55.0]
  HPV-18 [at Month 24] (N=170;154) | 140.8 [123.8 to 160.2] | 55.0 [55.0 to 55.0]
  HPV-18 [at Month 30] (N=17;19) | 89.5 [67.6 to 118.7] | 55.0 [55.0 to 55.0]
  HPV-18 [at Month 36] (N=167;145) | 107.9 [96.0 to 121.2] | 55.0 [55.0 to 55.0]
  HPV-18 [at Month 42] (N=25;19) | 103.3 [80.3 to 132.9] | 55.0 [55.0 to 55.0]
  HPV-18 [at Month 48 (N=179;150) | 96.9 [87.7 to 107.0] | 56.7 [54.0 to 59.6]

9. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as pain that prevented normal everyday activities as assessed by inability to attend work or school and which necessitated the administration of corrective therapy. Grade 3 redness and swelling was defined as redness/swelling above 50 millimeter (mm).
Time Frame: Within 60 minutes after vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects with at least 1 vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 3730 | 3740
Subjects
  Any pain | 1627 | 1610
  Grade 3 pain | 25 | 20
  Any redness | 544 | 501
  Grade 3 redness > 50 mm | 0 | 2
  Any swelling | 207 | 201
  Grade 3 swelling > 50 mm | 0 | 1

10. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited General Symptoms.
Description: Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal, headache, myalgia, rash, urticaria and fever (Fever = oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)). Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal everyday activities as assessed by inability to attend work or school and which necessitated the administration of corrective therapy.Grade 3 urticaria = urticaria distributed on at least 4 body areas. Grade 3 fever = oral temperature > 39.0°C.
Time Frame: Within 60 minutes after vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects with at least 1 vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 3730 | 3740
Subjects
  Any fatigue | 512 | 502
  Grade 3 fatigue | 6 | 5
  Any myalgia | 257 | 232
  Grade 3 myalgia | 0 | 1
  Any arthralgia | 58 | 64
  Grade 3 arthralgia | 0 | 1
  Any gastrointestinal | 191 | 171
  Grade 3 gastrointestinal | 0 | 0
  Any headache | 714 | 718
  Grade 3 headache | 2 | 0
  Any rash | 15 | 17
  Grade 3 rash | 0 | 0
  Any urticaria | 19 | 21
  Grade 3 urticaria | 0 | 0
  Fever (oral) >= 37.5°C | 472 | 477
  Fever (oral) > 39.0°C | 0 | 0

11. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms on a 10% Random Subset of Participants.
Description: as for outcome 9
Time Frame: From Day 3 to Day 6 after vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects with at least 1 vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 380 | 376
Subjects
  Any pain | 202 | 74
  Grade 3 pain | 0 | 0
  Any redness | 6 | 1
  Grade 3 redness | 1 | 0
  Any swelling | 23 | 1
  Grade 3 swelling | 7 | 0

12. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited General Symptoms on a 10% Random Subset of Participants.
Description: as for outcome 10
Time Frame: From Day 3 to Day 6 after vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects with at least 1 vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 380 | 376
Subjects
  Any pain | 214 | 189
  Grade 3 pain | 2 | 0
  Any myalgia | 250 | 211
  Grade 3 myalgia | 1 | 0
  Any arthralgia | 44 | 32
  Grade 3 arthralgia | 0 | 0
  Any gastrointestinal | 157 | 119
  Grade 3 gastrointestinal | 0 | 1
  Any headache | 247 | 242
  Grade 3 headache | 1 | 2
  Any rash | 31 | 26
  Grade 3 rash | 0 | 0
  Any urticaria | 3 | 1
  Grade 3 urticaria | 0 | 0
  Fever (oral) >= 37.5°C | 43 | 37
  Fever (oral) > 39.0°C | 0 | 0

13. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: During the entire study period (From Month 0 up to Month 48).
Population: The Total Vaccinated cohort included all vaccinated subjects with at least 1 vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 3727 | 3739
Subjects | 912 | 891

14. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs).
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the entire study period (From Month 0 up to Month 48).
Population: The Total Vaccinated cohort included all vaccinated subjects with at least 1 vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 3727 | 3739
Subjects | 3228 | 3254

15. Secondary Outcome: Number of Subjects With All Possible Pregnancy Outcomes
Description: The range of possible pregnancy outcomes was: Pregnancy loss, Pregnancy resolved alive, and Unresolved pregnancy.
Time Frame: During the entire study period (From Month 0 up to Month 48).
Population: The analysis was performed on the Total Vaccinated Cohort, on all pregnant subjects.
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 2123 | 2129
subjects
  Pregnancy loss | 317 | 294
  Pregnancy resolved alive | 1756 | 1766
  Unresolved pregnancy | 50 | 69

16. Secondary Outcome: Number of Cervical Infection With HPV16 or HPV18.
Description: as for outcome 2
Time Frame: During the first year of follow-up period
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 2380 | 2420
Events
  HPV16 Cervical Infection (N=2242;2232) | 21 | 37
  HPV18 Cervical Infection (N=2330;2347) | 7 | 29
  HPV16 and/or 18 Cervical Infection (N=2380;2420) | 27 | 64

17. Secondary Outcome: Number of Cervical Infection With HPV16 or HPV18.
Description: as for outcome 2
Time Frame: During the second year of follow-up period
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 2313 | 2349
Events
  HPV16 Cervical Infection (N=2170;2176) | 10 | 77
  HPV18 Cervical Infection (N=2269;2307) | 9 | 47
  HPV16 and/or 18 Cervical Infection (N=2313;2349) | 18 | 117

18. Secondary Outcome: Number of Cervical Infection With HPV16 or HPV18.
Description: as for outcome 2
Time Frame: During the third year of follow-up period
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 2232 | 2196
Events
  HPV16 Cervical Infection (N=2097;2026) | 6 | 60
  HPV18 Cervical Infection (N=2200;2196) | 6 | 44
  HPV16 and/or 18 Cervical Infection (N=2236;2166) | 11 | 88

19. Secondary Outcome: Number of Cervical Infection With HPV16 or HPV18.
Description: as for outcome 2
Time Frame: From the fourth year follow-up period
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 2421 | 2325
Events
  HPV16 Cervical Infection (N=2277;2139) | 13 | 77
  HPV18 Cervical Infection (N=2389;2325) | 10 | 57
  HPV16 and/or 18 Cervical Infection (N=2421;2261) | 22 | 118

20. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs).
Description: as for outcome 14
Time Frame: within 30 days (Days 0-29) after vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects with at least 1 vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Havrix Group
Number analyzed (Participants) | 3727 | 3739
Subjects | 1638 | 1536

ADVERSE EVENTS:
Time Frame: Solicited AEs: within 60 minutes after vaccination for all participants [please refer to Participant Flow Pre-assignment Details for population description]; From Day 3 to Day 6 post-vaccination for a 10% random subset of participants. SAEs: From Month 0 up to Month 48. Unsolicited AEs: From Month 0 up to Month 48 and Within 30 days (Days 0-29) after vaccination
Description: For this study, the Total Number (#) of Participants Affected by Other (non-serious) Adverse Events (AEs) was analyzed separately for expected AEs and for unexpected AEs. A consolidated analysis of all expected and unexpected AEs was not technically possible to be performed and the relevant data are no longer available. Therefore, the Total #Participants Affected in Other Adverse Events Table is currently populated by the highest value of #Participants affected within other AE's table.
Arm/Group | Cervarix Group | Havrix Group
Serious Adverse Events (participants affected / at risk) | 912/3727 | 891/3739
Other Adverse Events (participants affected / at risk) | 1627/3730 | 1610/3740
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=3727) | Havrix Group (N=3739)
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 134 | 108
False labour (Pregnancy, puerperium and perinatal conditions) | 66 | 88
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 64 | 64
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 59 | 63
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 57 | 64
Caesarean section (Surgical and medical procedures) | 56 | 59
Uterine hypotonus (Pregnancy, puerperium and perinatal conditions) | 54 | 54
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 39 | 53
Dengue fever (Infections and infestations) | 38 | 48
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 42 | 37
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 33 | 45
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 40 | 33
Urinary tract infection (Infections and infestations) | 25 | 24
Anaemia of pregnancy (Blood and lymphatic system disorders) | 24 | 22
Cholecystitis (Hepatobiliary disorders) | 26 | 19
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 18 | 23
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 19 | 20
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 18 | 19
Intentional self-injury (Psychiatric disorders) | 20 | 17
Appendicitis (Infections and infestations) | 17 | 18
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 16 | 18
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 18 | 14
Cholelithiasis (Hepatobiliary disorders) | 22 | 9
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 11 | 19
Obstructed labour (Pregnancy, puerperium and perinatal conditions) | 13 | 15
Abnormal product of conception (Pregnancy, puerperium and perinatal conditions) | 14 | 11
Postoperative wound infection (Infections and infestations) | 12 | 12
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 9 | 14
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 13 | 7
Postpartum sepsis (Infections and infestations) | 12 | 8
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 11 | 8
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 7
Gastrointestinal disorder (Gastrointestinal disorders) | 9 | 9
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 5 | 10
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 6 | 8
Multiple injuries (Injury, poisoning and procedural complications) | 3 | 10
Gestational diabetes (Metabolism and nutrition disorders) | 5 | 6
Hypertension (Vascular disorders) | 5 | 6
Ovarian cyst (Reproductive system and breast disorders) | 5 | 6
Pancreatitis acute (Gastrointestinal disorders) | 6 | 5
Multiple pregnancy (Pregnancy, puerperium and perinatal conditions) | 8 | 2
Placenta praevia haemorrhage (Pregnancy, puerperium and perinatal conditions) | 6 | 4
Subcutaneous abscess (Infections and infestations) | 5 | 5
Uterine haemorrhage (Reproductive system and breast disorders) | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 6 | 3
Foetal disorder (Pregnancy, puerperium and perinatal conditions) | 7 | 2
Depression (Psychiatric disorders) | 5 | 3
Infectious peritonitis (Infections and infestations) | 6 | 2
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 4 | 4
Mental disorder (Psychiatric disorders) | 5 | 3
Injury (Injury, poisoning and procedural complications) | 2 | 5
Menometrorrhagia (Reproductive system and breast disorders) | 5 | 2
Postoperative wound complication (Injury, poisoning and procedural complications) | 4 | 3
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 5 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 4
Pelvic inflammatory disease (Infections and infestations) | 3 | 3
Premature labour (Pregnancy, puerperium and perinatal conditions) | 2 | 4
Pyrexia (General disorders) | 5 | 1
Transverse presentation (Pregnancy, puerperium and perinatal conditions) | 3 | 3
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 4 | 1
Cardiovascular disorder (Cardiac disorders) | 5 | 0
Cellulitis (Infections and infestations) | 1 | 4
Concussion (Injury, poisoning and procedural complications) | 2 | 3
Essential hypertension (Vascular disorders) | 4 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 4
Salpingitis (Infections and infestations) | 3 | 2
Staphylococcal infection (Infections and infestations) | 3 | 2
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 3 | 2
Breast inflammation (Reproductive system and breast disorders) | 2 | 2
Bronchopneumonia (Infections and infestations) | 1 | 3
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 3
Endometriosis (Reproductive system and breast disorders) | 2 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 2
Open wound (Injury, poisoning and procedural complications) | 3 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 3
Perineal pain (Reproductive system and breast disorders) | 1 | 3
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 4 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1
Viral infection (Infections and infestations) | 1 | 3
Abortion complicated (Pregnancy, puerperium and perinatal conditions) | 3 | 0
Amniotic cavity infection (Infections and infestations) | 1 | 2
Bartholin's abscess (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 2 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 2
Circulatory collapse (Vascular disorders) | 2 | 1
Colitis ulcerative (Gastrointestinal disorders) | 2 | 1
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 0 | 3
Genital disorder female (Reproductive system and breast disorders) | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 3
Lymphadenitis (Blood and lymphatic system disorders) | 2 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 2
Migraine (Nervous system disorders) | 2 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Physical assault (Social circumstances) | 3 | 0
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Sexually transmitted disease (Infections and infestations) | 1 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Anaphylactic shock (Immune system disorders) | 0 | 2
Appendix disorder (Gastrointestinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 1 | 1
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Blood disorder (Blood and lymphatic system disorders) | 1 | 1
Cervix disorder (Reproductive system and breast disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Convulsion (Nervous system disorders) | 1 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 1
HIV infection (Infections and infestations) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Nervous system disorder (Nervous system disorders) | 0 | 2
Otitis externa (Infections and infestations) | 2 | 0
Parametritis (Infections and infestations) | 1 | 1
Phlebitis (Vascular disorders) | 0 | 2
Pneumonia (Infections and infestations) | 2 | 0
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 2
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 2 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 | 0
Tension headache (Nervous system disorders) | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0
Tooth abscess (Infections and infestations) | 2 | 0
Traumatic delivery (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 1
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Uterine polyp (Reproductive system and breast disorders) | 1 | 1
Vaginal infection (Infections and infestations) | 1 | 1
Varicose vein (Vascular disorders) | 0 | 2
Venom poisoning (Injury, poisoning and procedural complications) | 0 | 2
Abdominal mass (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abortion incomplete complicated (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Abortion spontaneous incomplete complicated (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary cirrhosis (Hepatobiliary disorders) | 1 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0
Breast abscess (Infections and infestations) | 1 | 0
Breast disorder (Reproductive system and breast disorders) | 1 | 0
Breast enlargement (Reproductive system and breast disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Candida sepsis (Infections and infestations) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Complicated migraine (Nervous system disorders) | 0 | 1
Congenital flat feet (Congenital, familial and genetic disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Drug dependence (Psychiatric disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Embolism venous (Vascular disorders) | 0 | 1
Emotional disorder (Psychiatric disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Eye complication associated with device (General disorders) | 1 | 0
Eye degenerative disorder (Eye disorders) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral hernia (Gastrointestinal disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Foetal malposition (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Genital herpes (Infections and infestations) | 1 | 0
Genitourinary tract infection (Infections and infestations) | 0 | 1
Granuloma skin (Skin and subcutaneous tissue disorders) | 0 | 1
Haematocolpos (Reproductive system and breast disorders) | 0 | 1
Haematosalpinx (Reproductive system and breast disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intracranial hypotension (Nervous system disorders) | 1 | 0
Intrapartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Malaria (Infections and infestations) | 1 | 0
Mastitis postpartum (Infections and infestations) | 0 | 1
Medical observation (Investigations) | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0
Multiple congenital abnormalities (Congenital, familial and genetic disorders) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Ovarian torsion (Reproductive system and breast disorders) | 0 | 1
Ovulation pain (Reproductive system and breast disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Pelvic haematoma obstetric (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0
Peritoneal disorder (Gastrointestinal disorders) | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0
Placental disorder (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Placental neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 1
Polymenorrhagia (Reproductive system and breast disorders) | 1 | 0
Post abortion haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Postpartum disorder (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Previous caesarean section (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Pyoderma (Infections and infestations) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Retinal disorder (Eye disorders) | 0 | 1
Rhesus incompatibility (Immune system disorders) | 0 | 1
Sexual abuse (Social circumstances) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Strabismus (Eye disorders) | 1 | 0
Syphilis (Infections and infestations) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Therapeutic procedure (Surgical and medical procedures) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Tooth ankylosis (Gastrointestinal disorders) | 1 | 0
Tooth development disorder (Gastrointestinal disorders) | 1 | 0
Tooth malformation (Gastrointestinal disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Twin pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0
Uterine inversion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Varicella (Infections and infestations) | 0 | 1
Varicophlebitis (Vascular disorders) | 0 | 1
Vascular headache (Nervous system disorders) | 1 | 0
Vulval abscess (Infections and infestations) | 1 | 0
Vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cervarix Group (N=3730) | Havrix Group (N=3740)
Pain (General disorders) | 1627 | 1610 — Within 60 minutes after vaccination.
Redness (General disorders) | 544 | 501 — Within 60 minutes after vaccination.
Swelling (General disorders) | 207 | 201 — Within 60 minutes after vaccination.
Fatigue (General disorders) | 512 | 502 — Within 60 minutes after vaccination.
Myalgia (General disorders) | 257 | 232 — Within 60 minutes after vaccination.
Gastrointestinal (General disorders) | 191 | 171 — Within 60 minutes after vaccination.
Headache (General disorders) | 714 | 718 — Within 60 minutes after vaccination.
Fever (General disorders) | 472 | 477 — Within 60 minutes after vaccination.
Pain (General disorders) | 202/380 | 74/376 — From Day 3 to Day 6 post-vaccination, in a 10% random subset of participants.
Swelling (General disorders) | 23/380 | 1/376 — From Day 3 to Day 6 post-vaccination, in a 10% random subset of participants.
Fatigue (General disorders) | 214/380 | 189/376 — From Day 3 to Day 6 post-vaccination, in a 10% random subset of participants.
Myalgia (General disorders) | 250/380 | 211/376 — From Day 3 to Day 6 post-vaccination, in a 10% random subset of participants.
Arthralgia (General disorders) | 44/380 | 32/376 — From Day 3 to Day 6 post-vaccination, in a 10% random subset of participants.
Gastrointestinal (General disorders) | 157/380 | 119/376 — From Day 3 to Day 6 post-vaccination, in a 10% random subset of participants.
Headache (General disorders) | 247/380 | 242/376 — From Day 3 to Day 6 post-vaccination, in a 10% random subset of participants.
Rash (General disorders) | 31/380 | 26/376 — From Day 3 to Day 6 post-vaccination, in a 10% random subset of participants.
Fever (General disorders) | 43/380 | 37/376 — From Day 3 to Day 6 post-vaccination, in a 10% random subset of participants.
Influenza (Infections and infestations) | 263/3727 | 293/3739 — Within 30 days (Days 0-29) after vaccination
Myalgia (Musculoskeletal and connective tissue disorders) | 355/3727 | 166/3739 — Within 30 days (Days 0-29) after vaccination
Headache (Nervous system disorders) | 218/3727 | 214/3739 — Within 30 days (Days 0-29) after vaccination
Menstruation irregular (Reproductive system and breast disorders) | 1021/3727 | 1011/3739 — From Month 0 up to Month 48
Influenza (Infections and infestations) | 903/3727 | 950/3739 — From Month 0 up to Month 48
Vaginal infection (Infections and infestations) | 709/3727 | 763/3739 — From Month 0 up to Month 48
Vulvovaginal candidiasis (Infections and infestations) | 714/3727 | 678/3739 — From Month 0 up to Month 48
Urinary tract infection (Infections and infestations) | 555/3727 | 565/3739 — From Month 0 up to Month 48
Upper respiratory tract infection (Infections and infestations) | 324/3727 | 327/3739 — From Month 0 up to Month 48
Headache (Nervous system disorders) | 324/3727 | 315/3739 — From Month 0 up to Month 48
Myalgia (Musculoskeletal and connective tissue disorders) | 386/3727 | 189/3739 — From Month 0 up to Month 48
Gastrointestinal inflammation (Gastrointestinal disorders) | 263/3727 | 249/3739 — From Month 0 up to Month 48
Dengue fever (Infections and infestations) | 174/3727 | 190/3739 — From Month 0 up to Month 48

LIMITATIONS AND CAVEATS:
The following analysis "occurence of histopathologically confirmed CIN2+ cases associated with HPV16 or HPV18 infection was not performed, in accordance with the Statistical Analysis Plan submitted to the FDA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.